CLINICAL TRIAL: NCT01762696
Title: A Real-time, Contextual Intervention Using PDAs to Reduce Marijuana Use in Youth
Brief Title: A Real-time, Contextual Intervention Using Mobile Technology to Reduce Marijuana Use in Youth
Acronym: MOMENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Lydia Shrier, Attending Physician, Adolescent Medicine, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R34DA030535-01A1 (NIH)
Record Dates: First submitted 2013-01-04; First posted 2013-01-08 (Estimated); Last update posted 2016-12-12 (Estimated); Status verified 2016-12

CONDITIONS: Marijuana Abuse
Keywords: marijuana; intervention; adolescent, young adult; primary care; mobile
MeSH Terms: conditions — Marijuana Abuse | interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MET only (Active Comparator): Motivational Enhancement Therapy only
  Interventions: Behavioral: MET
- MOMENT (Experimental): The full MOMENT intervention: Motivational Enhancement Therapy + momentary and daily mobile self-monitoring + motivational feedback messages prompting participants to consider their individualized coping strategies to avoid using marijuana
  Interventions: Behavioral: MET; Behavioral: MOMENT

INTERVENTIONS:
Behavioral: MET — Motivational Enhancement Therapy only
  Other Names: Motivational Enhancement Therapy
Behavioral: MOMENT — The full MOMENT intervention: Motivational Enhancement Therapy + momentary and daily mobile self-monitoring + motivational feedback messages prompting participants to consider their individualized coping strategies to avoid using marijuana
  Arms: MOMENT

SUMMARY:
The purpose of this study is to further develop and test the Momentary Self-Monitoring and Feedback + Motivational Enhancement Therapy (MOMENT) intervention, a real-time, contextual intervention to reduce marijuana use among primary care patients.

DETAILED DESCRIPTION:
This study proposes a pilot randomized trial to further develop and test the Momentary Self-Monitoring and Feedback + Motivational Enhancement Therapy (MOMENT) intervention, a real-time, contextual intervention to reduce marijuana use over three months in 15-to-24-year-old primary care patients who use frequently. We will randomize youth to one of two arms (goal 30 per arm completing 3-month follow-up): 1) MOMENT (MET + momentary self-monitoring + context-dependent feedback), or 2) MET-only. The two study arms will permit evaluation of the contributions of the self-monitoring and feedback components of the intervention above-and-beyond the MET and directly test the influence of the intervention on the link between momentary context and marijuana-related outcomes.

The specific aims of the study are

Specific Aim 1: Continued Feasibility Evaluation. In our preliminary work, we demonstrated that 1) youth perceive MOMENT to be easy to understand, comfortable, motivating, and helpful in reducing their marijuana use, 2) we can recruit 4 participants/month (minimum rate for the proposed study), and 3) we can successfully implement a MOMENT intervention study in the proposed recruitment sites. Based on this work, we have identified additional areas of feasibility on which to focus in the proposed study. Specifically, we aim to achieve:

1a. A signal response rate of at least 70% during each of three periods of momentary data collection - baseline, intervention, and 3-month follow-up.

1b. A diary response rate of at least 70% during each momentary data collection period

1. c. A retention rate of at least 80% of participants at the 3-month follow-up.

   Specific Aim 2. Early-Stage Efficacy Exploration. Our preliminary work showed that both momentary and individual-level outcomes improved from baseline to three months post-intervention. The primary momentary outcomes are desire to use marijuana when in a triggering context and likelihood of use following exposure to a triggering context. The primary individual-level outcomes are number of use events/week, 30-day percent of days abstinent, dose/use event, and measures of motivation (importance of, readiness for, and confidence about reducing use). Based on the preliminary findings, we will explore these early-stage efficacy questions:
2. a. Will improvements in momentary outcomes be observed with MOMENT, but not MET-only?

(1) The association between exposure to self-identified trigger contexts and momentary desire to use marijuana will be attenuated at three months, compared to pre-intervention.

(2) The likelihood of marijuana use following exposure to a trigger context will be reduced at three months.

2b. Will improvements in individual-level outcomes be greater with MOMENT vs. MET-only?

1. The reduction in marijuana use frequency (events/week and 30-day percent of days abstinent) and dose (per use event) will be greater at three months.
2. The increase in motivation to reduce or discontinue use will be greater at three months.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between the ages of 15-24 years
* Patient of the Boston Children's Hospital Adolescent/Young Adult Medicine Clinic or Martha Elliot Health Center Adolescent Clinic
* Ability to read and understand English

Exclusion Criteria:

* Medically or emotionally unstable, intoxicated or "high,", or otherwise unable to give consent at the time of their appointment
* Have previously participated in this study
* Does not meet the above inclusion criteria

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Actual)
Dates: Start 2013-05; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Marijuana desire | 3 months
  Desire to use marijuana when in top-3 trigger context
Marijuana use following trigger exposure | 3 months
  Marijuana use following exposure to top-3 trigger context
Frequency of marijuana use | 3 months
  Marijuana use events/day
Percent days abstinent | 3 months
  30-day percent days abstinent from marijuana use
Motivation to reduce marijuana use | 3 months
  Daily score on 3 scales - readiness to reduce marijuana use, importance of reducing use, and confidence in ability to reduce use

CONTACTS AND LOCATIONS:
Overall Officials: Lydia A Shrier, MD, MPH, Principal Investigator — Boston Children's Hospital
Locations (2):
- United States (2):
  - Boston Children's Hospital Adolescent/Young Adult Medical Clinic, Boston, Massachusetts
  - Martha Eliot Health Center Adolescent Clinic, Jamaica Plain, Massachusetts

REFERENCES:
- [Derived] Shrier LA, Harris SK. Associations of Momentary Mindfulness With Affect and Cannabis Desire in a Trial of Cannabis Use Interventions With and Without Momentary Assessment. J Adolesc Health. 2023 Jan;72(1):126-129. doi: 10.1016/j.jadohealth.2022.09.002. Epub 2022 Oct 20. PMID 36272891